CLINICAL TRIAL: NCT00344630
Title: TC-WYRE: TAXUS Express Stent vs. Cypher Stent - What's Your Real Life Experience?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: S5572; BSC
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: TAXUS Stent and Cypher Stent

SUMMARY:
To compare the relative efficacy and safety of the TAXUS Express2 stents and the Cypher stents among a broad, unselected patient population treated in a nationwide, multi-center clinical registry representative of 'real-world,' contemporary clinical practice. A secondary objective is to examine performance of the two stents in pre-specified subgroup populations and examine regional and national patterns in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with a TAXUS Express2 stent or a Cypher stent between April 1, 2005 and June 30, 2005.

Exclusion Criteria:

* Simultaneous treatment with both TAXUS and Cypher stents during the index revascularization. Patients who have undergone previous target vessel(s), stenting procedure within 9 months of the index procedure will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500
Dates: Start 2006-05; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: William O'Neill, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States